CLINICAL TRIAL: NCT03049306
Title: Propranolol for Sleep Apnea Therapy
Acronym: ProSAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00113241; 1R03HL138068-01 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2017-02-10 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; CPAP; Propranolol; Metabolism
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Propranolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Subjects will be admitted to the clinical research unit. On the CPAP withdrawal nights, placebo of propranolol LA (Inderal ® LA) 80 mg will be administered orally at 6:30 PM, after dinner. Blood pressure will be measured before administration, at 10:30 PM, and 6:30 AM. They will sleep from 10:30 PM to 6:30 AM. During sleep blood will be sampled from an indwelling IV for measurement of FFA, glucose, insulin, and triglycerides. This arm will is crossed-over with active drug 1 week before or after this study night.
  Interventions: Drug: Propranolol Oral Tablet; Drug: Placebo Oral Tablet
- Propranolol Oral Tablet (Active Comparator): Subjects will be admitted to the clinical research unit. On the CPAP withdrawal nights, Propranolol LA (Inderal ® LA) 80 mg will be administered orally before sleep, at 6:30 PM, after dinner. Blood pressure will be measured before administration, at 10:30 PM, and 6:30 AM. They will sleep from 10:30 Pm to 6:30 AM. During sleep blood will be sampled from an indwelling IV for measurement of FFA, glucose, insulin, and triglycerides. This arm will be crossed-over to placebo 1 week later. This arm will is crossed-over with active drug 1 week before or after this study night.
  Interventions: Drug: Propranolol Oral Tablet; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Propranolol Oral Tablet — Patients will receive Propranolol LA 80 mg PO at 7 PM before sleep (on CPAP withdrawal nights only)
  Other Names: beta blocker
Drug: Placebo Oral Tablet — Patients will receive Placebo tablet at 7 PM before sleep (on CPAP withdrawal nights only)
  Other Names: placebo

SUMMARY:
The primary objective of this study is to test whether a beta blocker, propranolol, lowers the overnight heart rate sleep in obstructive sleep apnea (OSA) during CPAP withdrawal. The secondary objectives are to test whether propranolol influences sleep architecture, morning blood pressure, and vascular function including reactive hyperemia index (RHI) and a marker of arterial stiffness, augmentation index (AIX).

DETAILED DESCRIPTION:
The overnight heart rate is increased in patients with obstructive sleep apnea (OSA), reflecting excessive sympathetic nervous system activity which may lead to long-term adverse cardiovascular consequences. Propranolol is a non-selective beta blocker that is used for a variety of indications including hypertension and anxiety. In this study investigators will administer propranolol or placebo to patients with OSA before sleep. Investigators will examine the effect of drug on nocturnal heart rate, morning blood pressure, and vascular health outcomes

ELIGIBILITY:
Inclusion Criteria:

* History of OSA (AHI>20, >50% events obstructive)
* Accustomed to CPAP use, and willing to discontinue CPAP temporarily for the study.
* If the participant has already completed "Metabolic Impact of Intermittent CPAP" (NA_00086830), they must have exhibited a >10% increase in nocturnal FFA or glucose during CPAP

Exclusion Criteria:

* Cardiovascular risks

  * Decompensated congestive heart failure
  * Atrial fibrillation, sick sinus syndrome, 2nd or 3rd degree heart block, pacemaker implantation, Wolff-Parkinson-White Syndrome (if not known, will check on a screening EKG)
  * Uncontrolled hypertension > 170/110
  * History of postural hypotension.
  * Resting systolic pressure <90 or heart rate < 50 on screening visit
* Drug interactions - currently taking any of the following drugs. (Subjects on these medications are excluded from participation and will not have the drug in question discontinued for the purposes of participation in the study. )

  * Calcium channel blockers that reduce heart rate (diltiazem, verapamil, fendiline, gallopamil)
  * Sympatholytic drugs: any other beta blocker; clonidine, terazosin or doxazosin; reserpine
  * Anti-arrhythmic drugs: (e.g. amiodarone, sotalol, digoxin, quinidine, lidocaine, propafenone)
  * Coumadin (propranolol may prolong INR)
  * Drugs that Inhibit CYP2D6, CYP1A2, or CYP2C19: amiodarone, ciprofloxacin, cimetidine, delavirdine, fluconazole, fluoxetine, fluvoxamine, imipramine, isoniazid, paroxetine, quinidine, ritonavir, rizatriptan, teniposide, theophylline, tolbutamide, zileuton, zolmitriptan
  * Drugs that increase hepatic metabolism of propranolol: rifampin, ethanol, phenytoin, and phenobarbital
  * Neuroleptics/anxiolytics: (thioridazine, chlorpromazine - may increase propranolol level), haloperidol, valium
  * Illicit drugs such as cocaine or amphetamines.
* Other medical conditions

  * Sleep disorder other than OSA, including: restless leg syndrome, parasomnia, or narcolepsy.
  * Shift work or circadian rhythm disorder that is expected to prevent good sleep as scheduled in the protocol
  * Insulin-dependent diabetes mellitus
  * Myasthenia gravis
  * Pheochromocytoma
  * Uncontrolled bronchospastic lung disease such as asthma or chronic obstructive pulmonary disease (COPD)
  * Current smoking
  * Chronic renal or liver failure
  * Known pregnancy, by urine testing in women of child-bearing age; nursing mothers
  * Known hypersensitivity to any beta blocker
* History of falling asleep while driving, near miss
* High risk occupation (pilot, commercial driver) Hemoglobin < 10 g/dL on point of care screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a history of obstructive sleep apnea (OSA) who were accustomed to continuous positive airway pressure (CPAP) use were enrolled from the Johns Hopkins Sleep Disorders Center. Patients with arrhythmias or taking beta blockers were excluded, among other criteria.
Pre-assignment Details: 24 participants signed a consent form. 1 subject was lost to follow up after consent, leaving 23 participants who were randomized to placebo first (n=11) or propranolol first (n=12).
Groups:
- Placebo First, Then Propranolol: This is a crossover study comparing placebo to propranolol taken before sleep prior to CPAP withdrawal. This arm received placebo during the first intervention and propranolol during the second intervention.
- Propranolol First, Then Placebo: This is a crossover study comparing placebo to propranolol taken before sleep prior to CPAP withdrawal. This arm received propranolol during the first intervention and placebo during the second intervention.
Period: First Intervention (1 Night)
Arm/Group | Placebo First, Then Propranolol | Propranolol First, Then Placebo
Started | 11 | 12
Completed | 10 | 11
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Second Intervention (1 Night)
Arm/Group | Placebo First, Then Propranolol | Propranolol First, Then Placebo
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Propranolol | Propranolol First, Then Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9) | 52 (13) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Heart Rate (Beats/Min, BPM)
Description: Average overnight heart rate (10:30 PM to 06:30 AM)
Time Frame: 1 Night (approximately 4 hours post administration for each intervention), from 10:30 PM to 06:30 AM
Measure: Mean (Standard Deviation); unit: BPM
Groups:
- Placebo Oral Tablet: Subjects will be admitted to the clinical research unit. On the CPAP withdrawal nights, placebo of propranolol LA (Inderal ® LA) 80 mg will be administered orally at 6:30 PM, after dinner. Blood pressure will be measured before administration, at 10:30 PM, and 6:30 AM. They will sleep from 10:30 PM to 6:30 AM. During sleep blood will be sampled from an indwelling IV for measurement of free fatty acids (FFA), glucose, insulin, and triglycerides. This arm will is crossed-over with active drug 1 week before or after this study night.
  Propranolol Oral Tablet: Patients will receive Propranolol LA 80 mg PO at 7 PM before sleep (on CPAP withdrawal nights only)
  Placebo Oral Tablet: Patients will receive Placebo tablet at 7 PM before sleep (on CPAP withdrawal nights only)
Arm/Group | Placebo Oral Tablet | Propranolol Oral Tablet
Number analyzed (Participants) | 21 | 21
BPM | 64.1 (5.1) | 60.2 (4.4)

2. Secondary Outcome: Reactive Hyperemia Index (RHI)
Description: Reactive Hyperemia Index (RHI) is measured by assessing the change in pulse wave amplitude in the brachial artery before and after a period of occlusion (usually 5 minutes). RHI is unitless as it reflects the ratio of pulse wave amplitude after : before occlusion. A high RHI indicates good endothelial function (values >1.67) and healthy vascular reactivity, while a low RHI (values <1.67) suggest endothelial dysfunction, which may be a risk factor for cardiovascular disease.
Time Frame: The morning after each intervention at 7:00 AM (approximately 11.5 hours post administration for each intervention)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo Oral Tablet | Propranolol Oral Tablet
Number analyzed (Participants) | 21 | 21
Ratio | 2.04 (0.55) | 2.11 (0.49)

3. Secondary Outcome: Systolic Blood Pressure (mmHg)
Description: Measured in the morning (7 AM)
Time Frame: The morning after each intervention at 7:00 AM (approximately 11.5 hours post administration for each intervention)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Oral Tablet | Propranolol Oral Tablet
Number analyzed (Participants) | 21 | 21
mmHg | 131 (14) | 125 (15)

4. Secondary Outcome: Diastolic Blood Pressure (mmHg)
Description: Measured in the morning (7 AM)
Time Frame: The morning after each intervention at 7:00 AM (approximately 11.5 hours post administration for each intervention)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Oral Tablet | Propranolol Oral Tablet
Number analyzed (Participants) | 21 | 21
mmHg | 80 (9) | 76 (11)

5. Secondary Outcome: Augmentation Index (%)
Description: The Augmentation Index (AIx) is measured by analyzing the arterial pulse wave, which captures the pressure wave reflections in the arteries. A higher AIx indicates increased arterial stiffness and higher cardiovascular risk, while a lower AIx suggests more compliant, healthier arteries. AIx can theoretically range from negative values to over 100%, although clinical values usually are between -10% and +40%.
Time Frame: The morning after each intervention at 7:00 AM (approximately 11.5 hours post administration for each intervention)
Measure: Mean (Standard Deviation); unit: Percentage of arterial pulse pressure
Arm/Group | Placebo Oral Tablet | Propranolol Oral Tablet
Number analyzed (Participants) | 21 | 21
Percentage of arterial pulse pressure | 14 (19) | 21 (18)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Description: We screened for the presence of:
  1. Bradycardia during nursing assessments during each study visit
  2. Hypotension (systolic BP <90 mmHg) during any point during the visit by BP cuff
Arm/Group | Placebo Oral Tablet | Propranolol Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT03049306/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03049306/SAP_001.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT03049306/ICF_002.pdf